CLINICAL TRIAL: NCT01116024
Title: ATS 3f Enable(tm) Aortic Bioprosthesis, Model 6000
Acronym: Enable
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2005 Rev. 17-MAY-2007
Record Dates: First submitted 2010-04-08; First posted 2010-05-04 (Estimated); Results first posted 2016-12-05 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2017-10

CONDITIONS: Heart Valve Diseases
Keywords: Diseased Heart Valve, Replacement, Aortic
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 3f Enable Aortic Bioprosthesis Model 6000 (Experimental): Single arm study
  Interventions: Device: ATS 3f Enable Aortic Bioprosthesis Model 6000

INTERVENTIONS:
Device: ATS 3f Enable Aortic Bioprosthesis Model 6000 — Replacement Aortic Heart Valve

SUMMARY:
This is a prospective, non-randomized, multi-center study designed to evaluate safety and effectiveness of the ATS 3f Enable Aortic Bioprosthesis in a patient population undergoing isolated aortic valve replacement with or without concomitant procedures. The Enable Aortic Valve is an equine pericardial stented bioprosthesis.

DETAILED DESCRIPTION:
The ATS 3f Enable Aortic Bioprosthesis is intended for those patients whose prognosis without surgical replacement of the diseased natural valve is unacceptably poor in terms of survival and/or quality of life in the opinion of the attending physicians. For these patients, there are a number of widely accepted prosthetic heart valves in use.

ELIGIBILITY:
Inclusion Criteria:

* The patient requires isolated aortic valve replacement with or without concomitant procedures such as coronary artery bypass or another valve repair. (The three remaining valves must be of native tissue).
* The patient is geographically stable and willing to return to the implant site for follow-up visits.
* The patient has been adequately informed of risks and requirements and consent to his/her participation in the clinical study.
* If this patient is female and of childbearing potential, patient has a negative pregnancy test within seven (7) days prior to the study procedure.

Exclusion Criteria:

* The patient requires replacement of two or more valves.
* The patient is < 20 years of age.
* The patient has a non-cardiac major or progressive disease, which in the Investigator's experience produces an unacceptable increased risk to the patient, or results in a life expectancy of less than 24 months.
* The patient is an intravenous drug and/or alcohol abuser.
* The patient presents with active endocarditis or other systemic infection.
* The patient has had previous valve replacement surgery, including previous implant and then explant of the ATS 3f Enable Aortic Bioprosthesis (Model 6000) or placement of a rigid annuloplasty ring in the mitral position.
* The patient is participating in concomitant research studies of investigational products.
* The patient presents with dilatation of the ascending aorta, Marfan Syndrome, Ehlers-Danlos syndrome, cystic medial degeneration, or other condition causing the ascending aorta to be irregular in geometry or physiology as seen via preoperative imaging.
* The patient has chronic renal failure.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2006-05; Primary Completion 2010-12 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Vang, Study Director — Medtronic
Locations (10):
- Medical University of Vienna, Vienna, Austria
- Germany (4):
  - Johann Wolfgang Goethe University, Frankfurt
  - University Medical Center Freiburg, Freiburg im Breisgau
  - University Medical Center Kiel, Kiel
  - UKSH, Campus Lubeck, Lübeck
- Poland (2):
  - Medical University of Gdansk, Gdansk
  - Jagiellonian University, Krakow
- Switzerland (2):
  - Cardiac Surgery University Hospital Basel, Basel
  - Inselspital Bern, Bern
- John Radcliffe Hospital, Oxford, United Kingdom

REFERENCES:
- See also: Medtronic, Inc. Corporate Website — http://www.medtronic.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients who required an aortic valve replacement were considered for this study if they met study preoperative selection criteria.
  Of 173 subjects enrolled, a cohort of 148 subjects was implanted and left the operating room with the study valve. Only subjects who left the operating room with the device implanted were included in the analysis.
Groups:
- ATS 3f Enable Aortic Bioprosthesis Model 6000: ATS 3f Enable Aortic Bioprosthesis Model 6000 : Replacement Aortic Heart Valve
Period: Overall Study
Arm/Group | ATS 3f Enable Aortic Bioprosthesis Model 6000
Started | 148 (148 subjects left operating room with the device implanted and were included in the analysis.)
Completed | 96 (Patient Enrollment stop date)
Not Completed | 52

BASELINE CHARACTERISTICS:
Population: 173 subjects were enrolled in the study. Of the 173 subjects enrolled, a cohort of 148 subjects were implanted with, and left the operating room with, the Model 6000 valve. As per protocol, only subjects who left the operating room with the device implanted were followed and included in the analysis.
Groups:
- Aortic Valve Replacement: 3f Enable Aortic Bioprosthesis Model 6000
Arm/Group | Aortic Valve Replacement
Number analyzed (Participants) | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.0 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91
  Male | 57
Region of Enrollment [Number; unit: participants]
  Austria | 6
  Poland | 31
  United Kingdom | 6
  Switzerland | 38
  Germany | 67

OUTCOME MEASURES:

1. Primary Outcome: Thromboembolism/Thrombosis
Description: Valve related thromboembolism and valvular thrombosis.
  Thrombosis was defined as any thrombus attached to or near the study valve that interfered with valve function in the absence of infection. The results are reported as linearized rate (percentage of participants per patient-year)
Time Frame: Five Years
Measure: Number (95% Confidence Interval); unit: percentage of participants/patient-year
Groups:
- Enable I Model 6000 Valve: Replacement Aortic Heart Valve: Study is single-arm. All subjects analyzed received the Enable I Model 6000 Valve.
Arm/Group | Enable I Model 6000 Valve: Replacement Aortic Heart Valve
Number analyzed (Participants) | 148
percentage of participants/patient-year
  Late Thromboembolism | 0 [0 to 0]
  Non-Structural Valve Dysfunction | 2.7 [1.4 to 5.2]
  All PVL | 2.4 [1.2 to 4.8]
  Major Paravalvular Leak | 1.5 [0.6 to 3.6]
  Thrombosis | 0 [0 to 0]

2. Primary Outcome: Hemorrhage/Bleeding-Anticoagulant/Antiaggregant (All and Major)
Description: Any episode of internal or external bleeding in subjects receiving anticoagulant and/or antiaggregant therapy.
  Hemorrhage/Bleeding (No Anticoagulant/Antiaggregant):
  Any episode of internal or external bleeding in subjects not receiving anticoagulant and/or antiaggregant therapy.
  The results are reported as linearized rate (percentage of participants per patient-year).
Time Frame: Five Years
Measure: Number (95% Confidence Interval); unit: percentage of participants/patient-year
Groups:
- Enable I Model 6000 Valve: Study is single-arm. All subjects analyzed received the Enable I Model 6000 Valve.
Arm/Group | Enable I Model 6000 Valve
Number analyzed (Participants) | 148
percentage of participants/patient-year
  All Hemorrhage Bleeding | 1.5 [0.6 to 3.6]
  Major Hemorrhage | 1.5 [0.6 to 3.6]
  Major Hemorrhage Bleeding Anticoagulant | 0.9 [0.3 to 2.8]
  Major Hemorrhage Bleeding No Anticoagulant | 0.6 [0.1 to 2.4]

3. Primary Outcome: Paravalvular Leaks (All and Major)
Description: Paravalvular leak was defined as any evidence of leakage of blood around the prosthesis (between the sewing ring and native annulus). Major Paravalvular leak was defined as any evidence of leakage of blood around the prosthesis, i.e. between the sewing ring and native annulus that requires surgical intervention.
  The results are reported as linearized rate (percentage of participants per patient-year).
Time Frame: Five Years
Measure: Number (95% Confidence Interval); unit: percentage of participants/patient-year
Arm/Group | Enable I Model 6000 Valve
Number analyzed (Participants) | 148
percentage of participants/patient-year
  All paravalvular leak | 2.4 [1.2 to 4.8]
  Major paravalvular leak | 1.5 [0.6 to 3.6]

4. Primary Outcome: Endocarditis
Description: Endocarditis was defined in the protocol as any infection involving the study valve. Any structural/non-structural valvular dysfunction, thrombosis, or embolic event associated with study valve endocarditis was captured as endocarditis only.
  The results are reported as linearized rate (percentage of participants per patient-year).
Time Frame: Five Years
Measure: Number (95% Confidence Interval); unit: percentage of participants/patient-year
Arm/Group | Enable I Model 6000 Valve: Replacement Aortic Heart Valve
Number analyzed (Participants) | 148
percentage of participants/patient-year | 0.9 [0.3 to 2.8]

5. Primary Outcome: Hemolysis
Description: Blood data analysis was performed in order to identify whether particular complications and serious adverse events such as hemolysis occurred. Hemolysis in subjects with tissue valves - as evidenced by increased serum lactate dehydrogenase concentrations, decreased serum haptoglobin concentration, erythrocytopenia and reticulocytosis - is usually associated with paravalvular leakage or infection.
Time Frame: Five Years
Measure: Number; unit: participants
Arm/Group | Enable I Model 6000 Valve: Replacement Aortic Heart Valve
Number analyzed (Participants) | 148
participants | 2

6. Primary Outcome: Structural Valve Deterioration
Description: Structural deterioration was defined as any change in the study valve function which resulted from an intrinsic abnormality that caused stenosis or regurgitation.
  There were no cases of structural deterioration reported for the study.
  The results are reported as linearized rate (percentage of participants per patient-year).
Time Frame: Five Years
Measure: Number; unit: percentage of participants/patient-year
Arm/Group | Enable I Model 6000 Valve: Replacement Aortic Heart Valve
Number analyzed (Participants) | 148
percentage of participants/patient-year | 0

7. Primary Outcome: Non-Structural Dysfunction
Description: Any abnormality resulting in stenosis or regurgitation at the operated valve that is not intrinsic to the valve itself. Non-structural dysfunction refers to non-structural problems that result in dysfunction of an operated valve exclusive of thrombosis and infection diagnosed by reoperation, autopsy, or clinical investigation.
  The results are reported as linearized rate (percentage of participants per patient-year).
Time Frame: Five Years
Measure: Number (95% Confidence Interval); unit: percentage of participants/patient-year
Arm/Group | Enable I Model 6000 Valve: Replacement Aortic Heart Valve
Number analyzed (Participants) | 148
percentage of participants/patient-year | 2.7 [1.4 to 5.2]

8. Primary Outcome: Re-operation, Explant, Repair
Description: Reoperation was defined in the protocol as any operation to repair, alter, or replace the study valve. Included is reoperation for repair of paravalvular leak and explant.
  The results are reported as linearized rate (percentage of participants per patient-year).
Time Frame: Five Years
Measure: Number (95% Confidence Interval); unit: percentage of participants/patient-year
Arm/Group | Enable I Model 6000 Valve: Replacement Aortic Heart Valve
Number analyzed (Participants) | 148
percentage of participants/patient-year
  Reoperation (All) | 2.1 [1.0 to 4.4]
  Explant | 2.1 [1.0 to 4.4]
  Repair | 0 [0 to 0]

9. Primary Outcome: Effectiveness Endpoint - NYHA Classification, Hemodynamic Performance
Description: New York Heart Association (NYHA) classification to asses improvement of the cardiac status, Hemodynamic Performance analysis based on Doppler echocardiographic studies.
  Class I: Patients with cardiac disease but without limitations of ordinary activity.
  Class II: Patients with cardiac disease resulting in slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea or anginal pain.
  Class III: Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary physical activity results in fatigue, palpitations or anginal pain.
  Class IV: Patients with cardiac disease resulting in inability to carry out any physical activity without discomfort. Symptoms of cardiac insufficiency or anginal syndrome may be present even at rest. If any physical activity is undertaken discomfort is increased.
Time Frame: Five Years
Measure: Number; unit: participants
Groups:
- NYHA Class Preoperative: Preoperative numbers of NYHA classification.
- NYHA Class 3-6 Months: NYHA classification after 3-6 months.
- NYHA Class 11-14 Months: NYHA classification after 11-14 months.
- NYHA Class 2 Year: NYHA classification after 2 years.
- NYHA Class 3 Year: NYHA classification after 3 years.
- NYHA Class 4 Year: NYHA classification after 4 years.
- NYHA Class 5 Year: NYHA classification after 5 years.
Arm/Group | NYHA Class Preoperative | NYHA Class 3-6 Months | NYHA Class 11-14 Months | NYHA Class 2 Year | NYHA Class 3 Year | NYHA Class 4 Year | NYHA Class 5 Year
Number analyzed (Participants) | 148 | 119 | 109 | 93 | 71 | 32 | 3
participants
  Class I | 9 | 47 | 51 | 41 | 37 | 10 | 1
  Class II | 38 | 61 | 53 | 48 | 29 | 19 | 2
  Class III | 92 | 4 | 4 | 4 | 5 | 3 | 0
  Class IV | 3 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown | 6 | 7 | 1 | 0 | 0 | 0 | 0

10. Primary Outcome: Hemodynamic
Description: Mean and peak pressure gradients from discharge through 5 years follow up. The gradient represents the difference in blood pressure across the valve.
Time Frame: Five Years
Population: At discharge, gradient data was collected of 103 subjects.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Discharge: Gradient at discharge
- 3-6 Months: Gradient at 3-6 Months
- 11-14 Months: Gradient at 11-14 months
- 2 Years: Gradient at 2 Years
- 3 Years: Gradient at 3 Years
- 4 Years: Gradient at 4 Years
- 5 Years: Gradient at 5 Years
Arm/Group | Discharge | 3-6 Months | 11-14 Months | 2 Years | 3 Years | 4 Years | 5 Years
Number analyzed (Participants) | 103 | 98 | 89 | 74 | 62 | 42 | 2
mmHg
  Mean Gradient | 10.28 (4.37) | 9.02 (3.70) | 8.59 (3.19) | 8.52 (3.39) | 8.77 (4.37) | 8.53 (4.79) | 5.55 (1.20)
  Peak Gradient | 20.38 (8.40) | 18.15 (7.17) | 16.58 (6.16) | 16.65 (6.89) | 17.69 (8.77) | 17.04 (8.75) | 10.30 (3.54)

11. Primary Outcome: Hemodynamics - Effective Orifice Area
Description: Effective orifice area (EOA) data.
  The effective orifice area is a measure of how much the heart valve prosthesis impedes blood flow through the aortic valve.
Time Frame: Five Years
Population: At discharge Effective Orifice Area data was collected for 61 subjects.
Measure: Mean (Standard Deviation); unit: EOA (cm2)
Groups:
- Discharge: Effective Orifice Area at discharge
- 3-6 Months: Effective Orifice Area at 3-6 months
- 11-14 Months: Effective Orifice Area at 11-14 months
- 2 Years: Effective Orifice Area at 2 years
- 3 Years: Effective Orifice Area at 3 years
- 4 Years: Effective Orifice Area at 4 years
- 5 Years: Effective Orifice Area at 5 years
Arm/Group | Discharge | 3-6 Months | 11-14 Months | 2 Years | 3 Years | 4 Years | 5 Years
Number analyzed (Participants) | 61 | 73 | 66 | 51 | 44 | 34 | 2
EOA (cm2) | 1.71 (0.45) | 1.68 (0.51) | 1.70 (0.46) | 1.66 (0.47) | 1.67 (0.43) | 1.62 (0.41) | 1.75 (0.0)

12. Primary Outcome: Hemodynamics - Effective Orifice Area Index
Description: The effective orifice area index is a measure of how much the heart valve prosthesis impedes blood flow through the aortic valve.
Time Frame: Five Years
Population: At discharge Effective Orifice Area index data was collected for 61 subjects.
Measure: Mean (Standard Deviation); unit: EOAi (cm2/m2)
Arm/Group | Discharge | 3-6 Months | 11-14 Months | 2 Years | 3 Years | 4 Years | 5 Years
Number analyzed (Participants) | 61 | 73 | 66 | 51 | 44 | 34 | 2
EOAi (cm2/m2) | 0.94 (0.25) | 0.91 (0.27) | 0.93 (0.25) | 0.89 (0.25) | 0.92 (0.25) | 0.89 (0.24) | 1.03 (0.06)

ADVERSE EVENTS:
Time Frame: 5 Years
Groups:
- Enable I Model 6000 Valve: Adverse events relating to the study safety endpoints.
Arm/Group | Enable I Model 6000 Valve
Serious Adverse Events (participants affected / at risk) | 39/148
Other Adverse Events (participants affected / at risk) | 3/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enable I Model 6000 Valve (N=148)
Valve-Related Adverse Event (Cardiac disorders) | 19 (19) — Seventeen out of 148 subjects (11.5%) experienced a Paravalvular Leak (PVL). Of these seventeen PVLs, nine events were reported as minor PVLs and eight events were reported as major PVLs. Three out of the 148 subjects (2.0%) developed endocarditis.
Not Valve-Related Adverse Event (Cardiac disorders) | 17 (17) — Five of the hemorrhage events were early events and three were late events.
Unknown Valve-Relatedness Adverse Event (Cardiac disorders) | 3 (3) — One out of the 148 subjects (0.7%) implanted experienced an early thromboembolism with a 21 mm valve. This subject experienced a peripheral arterial event, reported as unknown valve relatedness which resolved without permanent sequelae.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enable I Model 6000 Valve (N=148)
Unknown Valve Relatedness Adverse Event (Cardiac disorders) | 3 (3) — Unknown Valve Relatedness Adverse Event

LIMITATIONS AND CAVEATS:
Of the 173 subjects enrolled, a cohort of 148 subjects were implanted, followed and included in the analysis. 25 of the 173 subjects enrolled were intraoperative exclusions due to surgeon's discretion during the operative thoracotomy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No